CLINICAL TRIAL: NCT01361802
Title: A Multi-centre, Randomised, Double-blind, Placebo Controlled Parallel Group, Dose Finding Study to Assess the Efficacy and Safety of Ambroxol Spray (2.5mg, 5mg or 10mg) Versus Placebo for the Temporary Relief of Sore Throat Pain in Patients With Acute Pharyngitis
Brief Title: Ambroxol Spray Sore Throat Study
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 18.504
Record Dates: First submitted 2011-05-16; First posted 2011-05-27 (Estimated); Last update posted 2014-05-16 (Estimated); Status verified 2014-04

CONDITIONS: Pharyngitis; Pain
MeSH Terms: conditions — Pharyngitis; Pain

ARMS (4):
- Ambroxol Spray 2.5mg (Active Comparator): Ambroxol Spray Low Dose
  Interventions: Drug: Ambroxol Spray
- Ambroxol Spray 5mg (Active Comparator): Ambroxol Spray Medium Dose
  Interventions: Drug: Ambroxol Spray
- Ambroxol Spray 10mg (Active Comparator): Ambroxol Spray High dose
  Interventions: Drug: Ambroxol Spray
- Placebo Spray (Placebo Comparator): Placebo Spray
  Interventions: Drug: Placebo Spray

INTERVENTIONS:
Drug: Ambroxol Spray — low dose Ambroxol Spray
  Arms: Ambroxol Spray 2.5mg
Drug: Ambroxol Spray — medium dose Ambroxol Spray
  Arms: Ambroxol Spray 5mg
Drug: Ambroxol Spray — high dose Ambroxol Spray
  Arms: Ambroxol Spray 10mg
Drug: Placebo Spray — Placebo Spray
  Arms: Placebo Spray

SUMMARY:
The development of a new Ambroxol spray formulation for the treatment of sore throat pain associated with acute pharyngitis requires an initial phase II study to be conducted in order to select the most appropriate dose for pain relief.

ELIGIBILITY:
Inclusion criteria:

1. Sore throat due to acute pharyngitis (not more than 72 hours);
2. Score of 6 or greater on an 11-point pain intensity numerical rating scale;
3. Willingness to remain at the study centre for one hour following the first dose of study medication and return one to three days later.
4. Willing to take nothing by mouth except study medication for three hours following the first intake of study medication. Patients must also not smoke during this time period.

Exclusion criteria:

1. Known allergy to and/or hypersensitivity to ambroxol, sorbitol, or Acetaminophen;
2. Patients with drug dependence and/or alcohol abuse;
3. Use of any throat lozenge, throat spray, cough drop, menthol-containing product, or any product with demulcent properties within last 2 hours;
4. Use of any analgesic/anti-pyretic within last 4 hours;
5. Use of any "cold medication" (e.g. decongestant, antihistamine, expectorant, anti-tussive) within last eight hours;
6. Use of an antibiotic for an acute illness within last 24 hours;
7. Use of inhaled steroids or beta-agonists on a continuous basis during the last week;
8. Use of any investigational therapy (including a marketed drug taken for an investigational indication) within last 30 days
9. Any sign of mouth-breathing due to nasal congestion;
10. Cough that causes throat discomfort;
11. Active pulmonary disease such as bronchopneumonia;
12. Pregnant, lactating or breastfeeding women,
13. Any medical or psychiatric condition which, in the opinion of the investigator, could increase the risks associated with participation in an investigational study or affect compliance with the protocol.
14. Patients who have previously enrolled in this study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 494 (Actual)
Dates: Start 2011-05; Primary Completion 2011-08 (Actual)

PRIMARY OUTCOMES:
The primary endpoint is the time-weighted average of the pain intensity difference (PID) from pre-dose baseline over the first two hours after the first spray application expressed as a ratio of the pre-dose baseline (SPIDnorm0-2h). | 2 hours

SECONDARY OUTCOMES:
Patients will record their pain intensity on the 11-point ordinal numerical rating scale in the diary additionally at 3 hours after the first spray application and the corresponding SPIDnorm0-3h | 3 hours
Patients will record their pain intensity on the 11-point ordinal numerical rating scale in the diary additionally at 4, 6, 12 and 24 hours after the first spray application and the corresponding SPIDnorm0-24h | 4, 6, 12 and 24 hours
Patient assessment of efficacy at 3 and 24 hours after the first spray application will be assessed on a 5-point verbal rating scale. | 3 and 24 hours

CONTACTS AND LOCATIONS:
Overall Officials: Boehringer Ingelheim, Study Chair — Boehringer Ingelheim
Locations (15):
- South Africa (15):
  - 18.504.27015 Boehringer Ingelheim Investigational Site, Bloemfontein
  - 18.504.27005 Boehringer Ingelheim Investigational Site, Cape Town
  - 18.504.27011 Boehringer Ingelheim Investigational Site, Cape Town
  - 18.504.27013 Boehringer Ingelheim Investigational Site, Cape Town
  - 18.504.27014 Boehringer Ingelheim Investigational Site, Cape Town
  - 18.504.27008 Boehringer Ingelheim Investigational Site, Durban
  - 18.504.27010 Boehringer Ingelheim Investigational Site, Durban
  - 18.504.27001 Boehringer Ingelheim Investigational Site, Johannesburg
  - 18.504.27004 Boehringer Ingelheim Investigational Site, Klipspruit West
  - 18.504.27003 Boehringer Ingelheim Investigational Site, Krugersdorp
  - 18.504.27002 Boehringer Ingelheim Investigational Site, Lenasia
  - 18.504.27006 Boehringer Ingelheim Investigational Site, Newtown
  - 18.504.27012 Boehringer Ingelheim Investigational Site, Paarl
  - 18.504.27007 Boehringer Ingelheim Investigational Site, Pretoria
  - 18.504.27009 Boehringer Ingelheim Investigational Site, Sydenham